CLINICAL TRIAL: NCT01921582
Title: A Randomized Comparison of Osmotic Release Oral System Methylphenidate and Cognitive Behavioural Therapy for the Treatment of Obese Patients With Binge Eating Disorder
Brief Title: A Comparison of Methylphenidate and Cognitive Behavioural Therapy for the Treatment of Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Lena Quilty, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 044/2013
Record Dates: First submitted 2013-08-07; First posted 2013-08-13 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Methylphenidate; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate (TEVA-METHYLPHENIDATE ER-C)
  * Dosage: 18 mg/day at Week 1; 36 mg/day at Week 2; 54 mg/day at Week 3; 72 mg/day at Week 4. Dosage levels may be maintained or decreased to manage medication side effects.
  * Dosage form: tablet
  * Dosage frequency: daily
  * Duration: 12 weeks total
  Interventions: Drug: Methylphenidate
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy
  * 12 individual 50-minute appointments over the course of up to 14 weeks
  * According to Fairburn, Marcus, and Wilson (1993)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Methylphenidate — * Weekly appointments with study psychiatrists for the first four weeks, and then biweekly appointments for the last eight weeks.
  * Intervention will consist of medication as well as components of "Med-Plus" treatment (e.g., medication management, general support, and compliance enhancement strategies).
  Other Names: TEVA-METHYLPHENIDATE ER-C
  Arms: Methylphenidate
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavior Therapy will include three phases:
  * Phase 1 undertakes to eliminate binge episodes and introduce a 'regular' pattern of eating;
  * Phase 2 aims to reduce food intake and restructure eating-related cognitions;
  * Phase 3 focuses upon relapse prevention
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to determine whether methylphenidate is effective in the treatment of binge eating disorder, in a randomized controlled trial extended release methylphenidate versus cognitive behavioral therapy for binge eating disorder in overweight or obese adult females.

DETAILED DESCRIPTION:
Fifty-six adult female outpatients with binge eating disorder will receive 12 weeks of methylphenidate (dosage 18-72 mg) or 12 sessions of manualized cognitive behavioral therapy. Participants will complete interviewer-rated and self-report measures of eating, mood, attention, and personality features before treatment, after 6 weeks of treatment, immediately after treatment is completed, and 3 months after treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Binge-Eating Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
* Body Mass Index ≥ 25
* Must be fluent in English
* Must be capable to give informed consent

Exclusion Criteria:

* Current pregnancy or lactation
* Psychotherapy or behavioural treatment for eating or weight initiated during the past month
* Psychotropic or investigational medications initiated / changed during the past three months
* Concomitant use of another psychostimulant
* Current mental disorders that are acute/unstable, that require alternate treatment, and/or that preclude ability to complete research protocol including mania, psychosis, substance use (alcohol or drugs), dementia, organic brain disorders, mental retardation
* Current severe suicidality or homicidality
* Current uncontrolled medical conditions that affect weight or BED symptoms or that are contraindicated for methylphenidate including metabolic, neurological, hepatic, renal, cardiovascular, hematological, ophthalmic, or endocrine diseases
* Other serious medical illness or event such as acute myocardial infarction or stroke during the past six months
* History of seizures or tics in the past year
* Diagnosis or family history of Tourette's
* Clinically relevant laboratory results, including: Tachycardia as indicated by heart rate > 110; Hypertension as indicated by blood pressure parameters > 140 (systolic) and 90 (diastolic); Arrhythmias or conduction abnormalities as indicated by ECG parameters QTC> 460msec, QRS>120 msec, and PR>200 msec; Abnormal laboratory results (e.g., hypokalemia) as indicated by values > 20% above the upper range of the laboratory standard of a basic metabolic screen
* Current medications that affect weight
* Current medications that are contraindicated for methylphenidate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Frequency of binge episodes/days, as assessed by prospective daily binge diary | After 12 weeks of treatment

SECONDARY OUTCOMES:
Frequency of objective binge episodes and overall illness severity, as assessed by both the Eating Disorder Examination Interview and Questionnaire | After 12 weeks of treatment
Clinician impression of illness severity and improvement, as assessed by the Clinical Global Impression scale | After 12 weeks of treatment
Quality of life, as assessed by the Quality of Life Inventory | After 12 weeks of treatment
Associated features of binge eating as captured by the Dutch Eating Behavior Questionnaire and Binge Eating Scale | After 12 weeks of treatment
Body Mass Index | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lena C Quilty, PhD, Principal Investigator — Centre for Addiction and Mental Health; Allan S Kaplan, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research